CLINICAL TRIAL: NCT01507545
Title: A Randomized, Double-Blind, Placebo-controlled Study of the Efficacy & Safety of Monotherapy MORAb-004 Plus Best Supportive Care in Subjects With Chemorefractory Metastatic Colorectal Cancer
Brief Title: Morphotek Investigation in Colorectal Cancer: Research of MORAb-004 (MICRO)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: By the sponsor at the end of Stage 1 due to futility.
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MORAb-004-202-CRC
Record Dates: First submitted 2011-12-05; First posted 2012-01-11 (Estimated); Results first posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2015-09

CONDITIONS: Metastatic Colorectal Cancer; Colorectal Cancer
Keywords: mCRC; chemorefractory metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — ontuxizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MORAb-004 (Active Comparator)
  Interventions: Drug: MORAb-004; Other: Best supportive care
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Best supportive care

INTERVENTIONS:
Drug: MORAb-004 — MORAb-004 8mg per kg IV once a week
  Arms: MORAb-004
Drug: Placebo — Placebo - normal saline IV once a week
  Arms: Placebo
Other: Best supportive care — Best supportive care to improve quality of life

SUMMARY:
The purpose of this study is to evaluate whether therapy with MORAb-004 is effective and safe in the treatment of metastatic, colorectal cancer.

DETAILED DESCRIPTION:
Tumor endothelial marker-1 also referred to as TEM-1 is expressed in the supportive tissue, as well as, on the cells within the tumor. TEM-1, which is a cell surface glycoprotein, and is expressed in the stromal compartment (cells) of nearly all human tumors. In preclinical studies, it has been shown that TEM-1 plays a key role in tumor growth and the vascularization of tumors. There is evidence suggesting an association between the level of TEM-1, 7, 7R, 8 in relation to lymph node involvement and disease progression. MORAb-004 is a humanized immunoglobulin G (IgG1/κ) antibody directed against endosialin/TEM-1. Nonclinical pharmacological studies showed that MORAb-004 has the ability to block specific TEM-1 receptor-ligand interactions. Immunohistochemistry studies of human tumor biopsy samples demonstrate TEM-1 expression and MORAb-004 binding to tumor stromal cells, in particular mural cell compartment of neovessels and cancer-associated fibroblasts. All of which suggests a potential effective treatment. Researchers hypothesize that an antibody therapy that binds to TEM-1 may be efficacious in the treatment of metastatic, colorectal cancer. This clinical study is a proof of concept study to see if an anti-TEM-1 agent is safe and effective in the treatment of metastatic, colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >18 years old
* Diagnosis of metastatic, colorectal cancer
* Significant medical conditions must be well-controlled and stable for at least 30 days prior to the first treatment infusion
* Be willing and able to provide written informed consent

Exclusion Criteria:

* No prior treatment for metastatic colorectal cancer
* Other serious systemic diseases (bacterial or fungal)
* Clinically significant heart disease or an arrhythmia on an ECG within the past 6 months
* Known allergic reaction to monoclonal antibody therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-03-27 (Actual); Primary Completion 2013-10-20 (Actual); Study Completion 2013-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (66):
- United States (66):
  - Central Hem/Onc Medical Group, Inc., Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Providence St. Joseph Medical Center-Disney Family Cancer Center, Burbank, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - The Thomas and Dorothy Leavey Cancer Center Northridge Hospital Medical Center, Northridge, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - CPMCRI / Pacific Hematology Oncology Associates, San Francisco, California
  - Central Coast Medical Oncology, Santa Maria, California
  - UCLA Hematology Oncology, Santa Monica, California
  - Colorado Cancer Research Program, Denver, Colorado
  - St. Mary's Hospital Regional Cancer Center, Grand Junction, Colorado
  - Lutheran Hematology & Oncology, Wheat Ridge, Colorado
  - Christiana Care Health Services, Newark, Delaware
  - Georgetown University, Washington D.C., District of Columbia
  - Mayo Clinic Florida Hematology/Oncology, Jacksonville, Florida
  - Integrated Community Oncology Network / Cancer Specialists of North Florida, Jacksonville, Florida
  - Compass Research, LLC, Orange City, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Cancer Care Centers of Brevard, Rockledge, Florida
  - H. Lee Moffitt Cancer Center (Moffitt Cancer Center), Tampa, Florida
  - Suburban Hematology-Oncology Associates, P.C., Duluth, Georgia
  - Suburban Hematology-Oncology Assoc., PC, Lawrenceville, Georgia
  - Suburban Hematology-Oncology Associates, P.C., Snellville, Georgia
  - Medical and Surgical Specialists, Galesburg, Illinois
  - Ingalls Cancer Research Center, Harvey, Illinois
  - Oncology Specialists,S.C. Center for Advanced Care, Park Ridge, Illinois
  - Illinois CancerCare, P.C., Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Medical Oncology & Hematology Associates (Clinic #3), Clive, Iowa
  - Iowa Oncology Research Association, Des Moines, Iowa
  - Medical Oncology & Hematology Associates (Clinic #1), Des Moines, Iowa
  - Medical Oncology & Hematology Associates (Clinic #2), Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - John Hopkins University, Baltimore, Maryland
  - Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Essentia Health Duluth CCOP, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center/ CentraCare Health Plaza, Saint Cloud, Minnesota
  - Metro Minnesota CCOP, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Louis Park, Minnesota
  - St. John's Hospital, Saint Louis Park, Minnesota
  - CCCN, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Presbyterian Hospital Cancer Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Piedmont Hematology Oncology Associates PA, Winston-Salem, North Carolina
  - Medcenter One, Bismarck, North Dakota
  - TriHealth Oncology Institute/Oncology Partners Network, Cincinnati, Ohio
  - Hickman Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Cancer Center, Toledo, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Pharma Resource, East Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - St. Vincent Hospital / Green Bay Oncology, Green Bay, Wisconsin
  - St. Mary's Hospital / Green Bay Oncology, Green Bay, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 61 investigative sites in the United States from 27 March 2012 to 20 October 2013.
Pre-assignment Details: A total of 154 participants were screened and enrolled (signed informed consent form), of which 28 were screen failures, 126 were randomized and 122 were treated. Study was terminated by the sponsor at the end of Stage 1 due to futility, hence Stage 2 was not carried out.
Groups:
- MORAb-004 8.0 mg/kg + BSC: Participants received MORAb-004 8 milligram per kilogram (mg/kg), infusion intravenously (IV), once weekly, in each 2-week treatment cycle along with the best supportive care (BSC) which included those measures intended to provide palliation of all symptoms and improve quality of life, until disease progression or discontinuation from any reason (up to Cycle 24).
- Placebo + BSC: Participants received MORAb-004 matching placebo infusion IV, once weekly, in each 2-week treatment cycle along with the BSC which included those measures intended to provide palliation of all symptoms and improve quality of life, until disease progression or discontinuation from any reason (up to Cycle 24).
Period: Overall Study
Arm/Group | MORAb-004 8.0 mg/kg + BSC | Placebo + BSC
Started | 84 | 42
Treated/Safety Set | 82 | 40
Completed | 0 | 0
Not Completed | 84 | 42
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Discontinuation of the study by sponsor | 11 | 9
Not completed — Progressive disease | 60 | 27
Not completed — Other | 6 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants, analyzed according to the treatment assigned by the Interactive Voice Response System (IVRS) or Interactive Web Response System (IWRS).
Groups:
- MORAb-004 8.0 mg/kg + BSC: Participants received MORAb-004 8 mg/kg, infusion IV, once weekly, in each 2-week treatment cycle along with the BSC which included those measures intended to provide palliation of all symptoms and improve quality of life, until disease progression or discontinuation from any reason (up to Cycle 24).
- Total: Total of all reporting groups
Arm/Group | MORAb-004 8.0 mg/kg + BSC | Placebo + BSC | Total
Number analyzed (Participants) | 84 | 42 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (11.72) | 61.8 (10.61) | 61.5 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 16 | 59
  Male | 41 | 26 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 75 | 40 | 115
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 74 | 36 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS based on Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 was defined as the time (in weeks) from the date of randomization to the date of the first observation of disease progression (PD) or death due to any cause. PD was defined as at least a 20 percent (%) increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. If progression or death was not observed for a participant, the PFS time was censored at the date of last tumor assessment without evidence of progression prior to the date of initiation of further antitumor treatment. PFS was summarized for each treatment group using Kaplan-Meier estimation curves.
Time Frame: From the date of randomization to the date of the first observation of PD or death due to any cause (up to approximately 1 year 7 months)
Population: ITT population included all randomized participants, analyzed according to the treatment assigned by the IVRS/IWRS.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MORAb-004 8.0 mg/kg + BSC | Placebo + BSC
Number analyzed (Participants) | 84 | 42
weeks | 8.1 [7.9 to 8.1] | 8.1 [8.0 to 8.3]
Statistical Analysis 1: Comparison: MORAb-004 8.0 mg/kg + BSC vs Placebo + BSC; Test type: Superiority; p = 0.7335, One-sided log-rank test; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.76 to 1.67]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in months) from the date of randomization to the date of death, regardless of the cause. OS was summarized for each treatment group using Kaplan-Meier estimation curves. In the absence of death confirmation or for participants alive at the time of analysis, the survival time was censored at the last date known to be alive.
Time Frame: From the date of randomization to the date of death due to any cause (up to approximately 1 year 7 months)
Population: ITT population included all randomized participants, analyzed according to the treatment assigned by IVRS/IWRS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MORAb-004 8.0 mg/kg + BSC | Placebo + BSC
Number analyzed (Participants) | 84 | 42
months | 4.8 [3.7 to 6.2] | 6.2 [4.7 to 9.7]
Statistical Analysis 1: Comparison: MORAb-004 8.0 mg/kg + BSC vs Placebo + BSC; Test type: Superiority; p = 0.9498, One-sided log-rank test; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.93 to 2.19]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of subjects achieving either CR or PR using RECIST v.1.1. CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of randomization to the first documentation of CR or PR (up to approximately 1 year 7 months)
Population: ITT population included all randomized participants, analyzed according to the treatment assigned by IVRS/IWRS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MORAb-004 8.0 mg/kg + BSC | Placebo + BSC
Number analyzed (Participants) | 84 | 42
percentage of participants | 0 [0.000 to 4.296] | 2.4 [0.060 to 12.566]
Statistical Analysis 1: Comparison: MORAb-004 8.0 mg/kg + BSC vs Placebo + BSC; Test type: Superiority; p = 0.333, Fisher Exact; Difference of arms = -2.4, 95% CI 2-sided [-6.992 to 2.230]

4. Secondary Outcome: Time to Tumor Response (TTR)
Description: Time to tumor response was defined for those participants with objective evidence of confirmed CR or PR as the time from randomization to first documentation of objective tumor response (CR or PR). CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of randomization to first documentation of objective tumor response (CR or PR) (up to approximately 1 year 7 months)
Population: ITT population included all randomized participants, analyzed according to the treatment assigned by the IVRS/IWRS.
  Here overall number analyzed "N" are the participants who had achieved CR or PR.
Measure: Median (Full Range); unit: weeks
Arm/Group | MORAb-004 8.0 mg/kg + BSC | Placebo + BSC
Number analyzed (Participants) | 0 | 1
weeks |  | NA [NA to NA] — Data for TTR were not estimable because of low response rate (CR or PR) among all participants.

5. Secondary Outcome: Duration of Response (DOR)
Description: The DOR was defined as the time from first documentation of objective response (CR or PR) to the first documentation of objective tumor progression or death due to any cause. CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of first objective response (CR or PR) to objective tumor progression or death regardless of cause (up to approximately 1 year 7 months)
Population: as for outcome 4
Measure: Median (Full Range); unit: weeks
Arm/Group | MORAb-004 8.0 mg/kg + BSC | Placebo + BSC
Number analyzed (Participants) | 0 | 1
weeks |  | NA [NA to NA] — Data for DOR were not estimable because of low response rate (CR or PR) among all participants.

6. Secondary Outcome: Biomarkers Based PFS, Within Treatment Group
Description: The statistical evidence to support the use of the biomarker identified in Stage 1 interim analysis for Stage 2 selection of participants as designed was not adequate to clearly define a biomarker responsive population. The study was terminated by the sponsor at the end of Stage 1 and enrollment of stage 2 did not occur due to futility, hence Stage 2 and biomarker based analysis for PFS was not carried out.
Time Frame: From the date of randomization up to approximately 1 year 7 months
Population: The study was terminated by the sponsor at the end of Stage 1 and enrollment of stage 2 did not occur due to futility, hence Stage 2 and biomarker based analysis for PFS was not carried out.
Arm/Group | MORAb-004 8.0 mg/kg + BSC | Placebo + BSC
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Biomarkers Based OS, Within Treatment Group
Description: The statistical evidence to support the use of the biomarker identified in Stage 1 interim analysis for Stage 2 selection of participants as designed was not adequate to clearly define a biomarker responsive population. The study was terminated by the sponsor at the end of Stage 1 and enrollment of stage 2 did not occur due to futility, hence Stage 2 and biomarker based analysis for OS was not carried out.
Time Frame: From the date of randomization up to approximately 1 year 7 months
Population: The study was terminated by the sponsor at the end of Stage 1 and enrollment of stage 2 did not occur due to futility, hence Stage 2 and biomarker based analysis for OS was not carried out.
Arm/Group | MORAb-004 8.0 mg/kg + BSC | Placebo + BSC
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the date of randomization of the study drug up to 45 days after the last infusion of study drug (approximately up to 1 year 7 months)
Arm/Group | MORAb-004 8.0 mg/kg + BSC | Placebo + BSC
All-Cause Mortality (participants affected / at risk) | 13/82 | 4/40
Serious Adverse Events (participants affected / at risk) | 31/82 | 15/40
Other Adverse Events (participants affected / at risk) | 77/82 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MORAb-004 8.0 mg/kg + BSC (N=82) | Placebo + BSC (N=40)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 3 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Caecitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Gait Disturbance (General disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 3 | 0
Abdominal Wall Abscess (Infections and infestations) | 1 | 0
Intestinal Fistula Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Septic Shock (Infections and infestations) | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 2
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 2
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Cauda Equina Syndrome (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 2 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 2 | 1
Embolism (Vascular disorders) | 2 | 0
General Physical Health Deterioration (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MORAb-004 8.0 mg/kg + BSC (N=82) | Placebo + BSC (N=40)
Anaemia (Blood and lymphatic system disorders) | 10 | 5
Lymphopenia (Blood and lymphatic system disorders) | 6 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 4 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Sinus Arrhythmia (Cardiac disorders) | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Eye Pain (Eye disorders) | 1 | 0
Vision Blurred (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Eyelid Disorder (Eye disorders) | 0 | 1
Vitreous Floaters (Eye disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 32 | 14
Constipation (Gastrointestinal disorders) | 22 | 13
Abdominal Pain (Gastrointestinal disorders) | 16 | 8
Vomiting (Gastrointestinal disorders) | 17 | 9
Diarrhoea (Gastrointestinal disorders) | 16 | 6
Abdominal Distension (Gastrointestinal disorders) | 8 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 6 | 2
Ascites (Gastrointestinal disorders) | 5 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Faecal Volume Increased (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Lip Haematoma (Gastrointestinal disorders) | 1 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 2
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1
Gingival Pain (Gastrointestinal disorders) | 0 | 1
Perianal Erythema (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 43 | 19
Oedema Peripheral (General disorders) | 12 | 6
Pyrexia (General disorders) | 11 | 5
Asthenia (General disorders) | 8 | 4
Chills (General disorders) | 8 | 4
Pain (General disorders) | 7 | 0
Malaise (General disorders) | 4 | 0
Gait Disturbance (General disorders) | 3 | 0
Influenza Like Illness (General disorders) | 2 | 1
Non-Cardiac Chest Pain (General disorders) | 2 | 0
Early Satiety (General disorders) | 1 | 0
Injection Site Reaction (General disorders) | 1 | 0
Chest Discomfort (General disorders) | 0 | 1
Suprapubic Pain (General disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2
Drug Hypersensitivity (Immune system disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 8
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1
Abdominal Infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Diarrhoea Infectious (Infections and infestations) | 0 | 1
Oral Candidiasis (Infections and infestations) | 0 | 2
Oral Herpes (Infections and infestations) | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 10 | 1
Weight Decreased (Investigations) | 10 | 3
Aspartate Aminotransferase Increased (Investigations) | 6 | 1
Alanine Aminotransferase Increased (Investigations) | 5 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 5 | 4
Blood Bilirubin Increased (Investigations) | 3 | 0
Blood Creatinine Increased (Investigations) | 3 | 0
Electrocardiogram Abnormal (Investigations) | 3 | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2 | 2
Blood Cholesterol Increased (Investigations) | 1 | 0
Blood Magnesium Increased (Investigations) | 1 | 0
Blood Pressure Decreased (Investigations) | 1 | 0
Blood Uric Acid Increased (Investigations) | 1 | 1
Cardiac Murmur (Investigations) | 1 | 0
Ejection Fraction Decreased (Investigations) | 1 | 0
International Normalised Ratio Increased (Investigations) | 1 | 0
Lymphocyte Count Decreased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 0
Prothrombin Time Prolonged (Investigations) | 1 | 0
White Blood Cell Count Decreased (Investigations) | 1 | 0
Blood Glucose Increased (Investigations) | 0 | 1
Electrocardiogram ST Segment Depression (Investigations) | 0 | 1
Haemoglobin Decreased (Investigations) | 0 | 1
Peritoneal Fluid Analysis Abnormal (Investigations) | 0 | 1
Peritoneal Fluid Analysis Normal (Investigations) | 0 | 1
Transaminases Increased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 28 | 11
Dehydration (Metabolism and nutrition disorders) | 7 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Failure To Thrive (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Increased Appetite (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 15 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 9 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 7 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 16 | 8
Dizziness (Nervous system disorders) | 6 | 0
Neuropathy Peripheral (Nervous system disorders) | 3 | 3
Dysgeusia (Nervous system disorders) | 2 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 2 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 0
Brain Oedema (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Hypogeusia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 1
Memory Impairment (Nervous system disorders) | 1 | 0
Peroneal Nerve Palsy (Nervous system disorders) | 1 | 0
Restless Legs Syndrome (Nervous system disorders) | 1 | 1
Sinus Headache (Nervous system disorders) | 1 | 0
Slow Speech (Nervous system disorders) | 1 | 0
Balance Disorder (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 8 | 3
Anxiety (Psychiatric disorders) | 5 | 2
Depression (Psychiatric disorders) | 3 | 2
Libido Decreased (Psychiatric disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 5 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 2 | 2
Chromaturia (Renal and urinary disorders) | 1 | 0
Micturition Urgency (Renal and urinary disorders) | 1 | 0
Ureteric Stenosis (Renal and urinary disorders) | 1 | 0
Urinary Tract Pain (Renal and urinary disorders) | 1 | 1
Urine Flow Decreased (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 1
Nephrolithiasis 0 (Renal and urinary disorders) | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 1 | 1
Perineal Pain (Reproductive system and breast disorders) | 1 | 0
Scrotal Swelling (Reproductive system and breast disorders) | 1 | 0
Scrotal Pain (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 4 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Pain Of Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 6 | 3
Hypertension (Vascular disorders) | 5 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 0
Hot Flush (Vascular disorders) | 2 | 2
Haematoma (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated by the sponsor at the end of Stage 1 due to futility, hence Stage 2 was not carried out.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes